CLINICAL TRIAL: NCT02256163
Title: Identification of Genes and Pathogenesis Involved in Familial Thoracic Aortic Aneurysm (TAA)
Brief Title: Identification of Genes and Pathogenesis Involved in Familial Thoracic Aortic Aneurysm
Acronym: TAA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI10023; N° ID RCB: 2010-A01448-31 (Other: ANSM); AOM10108 (Other: AP-HP)
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Thoracic Aortic Aneurysm
Keywords: Thoracic Aortic Aneurysm (TAA); gene; familial TAA; blood collection
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample.
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objectives of the study are

* to assess the contribution of alteration of each known gene on non-syndromic TAA.
* to map and identify unknown gene involved in the non-syndromic TAA.

DETAILED DESCRIPTION:
The secondary objectives of the study are

* to study the correlation of phenotype-genotype, in particular, to compare the aortic phenotype of non-syndromic TAA patients and TAA syndromic patients.
* to develop national standardized strategies of genetic diagnosis and of clinical management using genetic data.

ELIGIBILITY:
Inclusion Criteria:

For all:

* Aged > 18 years.
* Written informed consent obtained.
* People with health insurance.

For individual:

* people ≥ 45 years, thoracic aortic aneurysm without syndrome,
* or people > 45 years with familial TAA.

For family:

* At least 2 members of family in 2 generations have TAA without syndrome and at least 2 patients of TAA will undergo blood collection.
* All people in family will undergo blood collection, each member should declare at first his (her) status (with or without TAA, unknown), the relationship (direct relative family or family in-law), no limit of age. For the children, only those with TAA will perform blood collection for the study.

Exclusion Criteria:

* Thoracic aortic aneurysm with different syndromes (Marfan syndrome, Ehlers-Danlos syndrome, Loeys-Dietz syndrome, Turner syndrome, Noonan syndrome).
* Arterial hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollement of individuals and families followed in the reference centers and the competence centers,
  * search for mutations in one of known genes such as FBN1, TGFBR1, TGFBR2, ACTA2, or MYH11.
  * search for new genes in families and individuals with TAA who without mutation in one of the known genes.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Impact of known mutations and research of new genes involved in non syndromic TAA | 1 year
  Research for mutations in known genes such as FBN1, TGFBR1, TGFBR2, ACTA2, or MYH11.
  Research for new genes in families and in individuals TAA patients without known mutation.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Boileau, MD, Principal Investigator — Département de Génétique, Hôpital Bichat, France
Locations (1):
- Département de Génétique, Hôpital Bichat, Paris, Île-de-France Region, France